CLINICAL TRIAL: NCT01421537
Title: Evaluation Of Enoxaparin Pharmacokinetic For Thromboprophylaxis In Burn Care Patients
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: CE 10.148
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Skin Burn Extensive
Keywords: Thromboprophylaxis; enoxaparin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
OVERVIEW:

* Thromboembolisms represent a serious and feared complication in hospitalized patients.
* Several factors make the ICU patient population at increased risk of venous thromboembolism.
* A high incidence of thromboembolic events is starting to emerge from recent medical literature in the burn patient.
* Actual guidelines for thromboprophylaxis in burn care patients are based on multiple non-burn patient trials.
* Burn patient physiology is radically different than that of general ward hospitalized patients
* Since the actual chemical thromboprophylaxis have not been evaluated in the burn patient, it is of interest to assess their efficacy in patients with severe burns.
* Hence, the pharmacokinetic characterization of heparins (a well accepted mode of thromboprophylaxis) in burn patients could guide future quality of care for this subclass of patients.

Our proposal is based on the conviction that anti-Xa activity of low-molecular-weight heparins in the burn patients do not correlate with levels described to prevent thromboembolic events in the general hospitalized population.

The investigators aim to:

1. To evaluate pharmacokinetics and pharmacodynamics of low-molecular-weight heparins (enoxaparin), with anti-Xa levels in severely burned patients receiving thromboprophylaxis.
2. To determine the correlation between antithrombotic activity of heparins and the different metabolic phases of the thermally injured patient.

DETAILED DESCRIPTION:
Deep venous thrombosis (DVT) has taken a prevalent place in medical literature over the past decades. In an attempt to decrease its impact on hospitalized patients, multiple trials have tried to better define its frequency and consequences on a very broad range of patients. The differences between these sub populations of ill individuals influence greatly the occurrence of venous thrombotic events (VTE).

Critically ill patients are predisposed to VTEs. The nature of the disease may have an important impact on the risk for DVT. Mechanical ventilation, central line placement, surgery, vasopressors and immobilization are some of the realities of ICU patients. They contribute to the enhanced chance for thromboembolic complications in this population, either by venous stasis (immobilization), endothelial injury (surgery…) or hypercoagulability. Trauma patients represent a subclass of critical care patients with a high incidence of DVT. It has been evaluated as high as 44,1% even in patients with thrombotic prophylaxis with low-dose unfractioned heparin.

Burn patient are also at increased risk of deep vein thrombosis and pulmonary embolisms. Recent prospective trials in burn patients have described an incidence of thromboembolic complications in the range of 6 to 60%. Autopsy evaluations are also in favor of an elevated incidence of thrombotic events in thermally injured patients(37 to 60%).

At the present time, no trial has evaluated the efficacy of the pharmacologic methods used for thromboprophylaxis in burned patients. Comparative efficacy between different patient populations (including thermally injured patients) has never been undertook. Thus, the investigators have to question the adequacy of present thromboprophylactic measures in burn patients? Are the actual method of DVT and PE prophylaxis sufficient in severe burns?

The physiology of moderate to severe burns makes us believe it is not. In the early post burn period, a massive fluid reanimation is initiated. The Starling forces are destabilized in favor of an increased capillary leak to the interstitial space. The net effect is the increase in free water in the interstitium and formation of important edema. The distance between the epithelium and the vascular space is then potentially increased. Furthermore, the central intravascular compartment of such individuals becomes very difficult to access. This leads us to reconsider the efficiency of the subcutaneous route. In cases of severe accumulation of interstitial fluid, can the subcutaneous administration of medications lead to the desired therapeutic effect?

The investigators plan to compare the levels of anti-Xa levels between 3 patient populations: severely burned patients (> 20%), medical ICU patients and general medical ward patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and over
* Burn injuries greater than 20%
* Received at least 24 hours of enoxaparin prior to the sampling series
* Patients admitted to Hôtel-Dieu hospital of the "CHUM: Centre hospitalier de l'Université de Montréal"

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Patients in the postoperative period (within 24 hours of the surgery)
* Patients with a contraindication for heparin use (Heparin induced thrombocytopenia and severe hemorrhage)
* Patients needing therapeutic anticoagulation
* Hepatic insufficiency prior to the burn injury (CHILD-PUGH B or more)
* Patients with a hemoglobin inferior to 70g/L
* Patients with a renal clearance less than 30 ml/min as calculated with the Cockroff-Gault formula prior to the burn care admission.
* Patients without basic French or English comprehension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients in :
  * general medical ward
  * mixte intensive care unit
  * burn patient intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Lafrance, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Anita Ang, M. Sc, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Nicholas Robillard, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Mikhael Laskine, MD, Principal Investigator — CHUM; Normand Blais, MD, Principal Investigator — CHUM; Sylvain Belisle, MD, Principal Investigator — CHUM; Marc-Jacques Dubois, MD, Principal Investigator — CHUM
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada